CLINICAL TRIAL: NCT03415243
Title: A Single Dose, Open Label, Randomized Scintigraphic Study to Investigate the Gastrointestinal Behavior of 2 Triple Combination Products (Acetaminophen, Phenylephrine and Dextromethorphan) in Healthy Male Volunteers
Brief Title: To Investigate the Gastrointestinal Behaviour of Two Triple Combination Products in Healthy Male Volunteers
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 208821
Record Dates: First submitted 2018-01-23; First posted 2018-01-30 (Actual); Results first posted 2019-06-24 (Actual); Last update posted 2019-06-24 (Actual); Status verified 2019-03

CONDITIONS: Common Cold
MeSH Terms: conditions — Common Cold | interventions — Acetaminophen; Dextromethorphan; Phenylephrine

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Treatment A Group (Experimental): Participants will receive a single dose (1 sachet) of the investigational product (Acetaminophen 650mg+Dextromethorphan 20mg+Phenylephrine 10mg).
  Interventions: Drug: Acetaminophen 650mg+Dextromethorphan 20mg+Phenylephrine 10mg
- Treatment B Group (Experimental): Participants will receive a single dose (2 caplets) of the investigational product (Acetaminophen 325mg+Dextromethorphan 10mg+Phenylephrine 5mg).
  Interventions: Drug: Acetaminophen 325mg+Dextromethorphan 10mg+Phenylephrine 5mg

INTERVENTIONS:
Drug: Acetaminophen 650mg+Dextromethorphan 20mg+Phenylephrine 10mg — Contents of the sachet will be emptied into a glass bottle and 225 mL of hot, but not boiling water (approximately 90-95°C), will be added to the container and mixed to dissolve the contents of the sachet. The dissolved solution will be allowed to cool to approximately 40 - 50 degree Celsius (°C). After cooling, a small volume (1 to 10 microliters [mcL]) of 99mTc-DTPA (Technetium-99m-diethylene-triamine-pentaacetate will be added to the drug solution in to achieve a maximum of 108 curie(mcCi) i.e.4 megabecquerel [MBq] per individual dose at the time of dosing. The container will be capped and maintained at a temperature between 35-45°C at time of dosing and then participants will be instructed to consume the hot drink entirely within 30 seconds.
  Other Names: Theraflu daytime severe cold and cough powder
  Arms: Treatment A Group
Drug: Acetaminophen 325mg+Dextromethorphan 10mg+Phenylephrine 5mg — Caplet doses will be prepared by drilling hole of approximately(app.)1millimetre(mm)diameter and app.2-2.5mm deep into individual caplets.99mTc-DTPA(dissolved in normal saline)will be added into hole of each caplet as low volume liquid(0.5-2.0mcL)to achieve maximum of 54 mcCi(2MBq)per caplet at time of dosing(2caplets=108 mcCi[4MBq]dose per assessment visit).Applied liquid will be allowed to air dry,hole to be filled with equivalent powder blend from crushed caplet so drug content will remain constant for all caplets.Caplet will be sealed with appropriate material.Radiolabeled caplets will be packaged as unit doses(2 caplets per container)and maintained at room temperature until administration.Caplets will be swallowed with 225mL of noncarbonated room temperature water within 30 seconds.
  Other Names: Theraflu expressmax daytime severe cold and cough caplets
  Arms: Treatment B Group

SUMMARY:
This clinical study will be conducted to characterize the gastrointestinal transit of two multi-symptoms formulations by inclusion of a radiolabel marker.

DETAILED DESCRIPTION:
This study will be an open label, randomized, single dose, parallel groups gamma scintigraphic study. A total of 28 healthy male participants will be randomized (14 participantper treatment arm) in order to have 24 evaluable participants (12 participants per treatment arm). Participants will be randomized to receive either a single dose Treatment A (Theraflu daytime Severe Cold & Cough powder) or single dose of Treatment B (Theraflu ExpressMax Daytime Severe Cold and Cough caplets). This study will consist of screening visit (Visit 1), followed by a treatment visit (Visit 2). Visit 2 includes two days: Day -1 and Day 1. On visit 2 (day -1) of the study, the study participants will be admitted to the unit at approximately 7 pm on the evening before study drug administration and will receive a standardized meal. Participants will be required to fast (nothing to eat or drink except non-carbonated water) from 10 hours prior until 4 hours after study drug administration. Water will be permitted until 1 hour prior to investigational product administration, and no additional fluids until the lunch meal will be served at approximately 4 hours post dose. Participants will then be given a standard lunch at 4 hours post-dose, a standard dinner at 10 hours post-dose on Day 1. Participants will be discharged from the unit after the last scintigraphic imaging is performed, blood sample for laboratory test will be taken as well as a brief physical examination. Scintigraphic acquisitions will be taken beginning after dose administration until 10 hours post-dose.

ELIGIBILITY:
Inclusion Criteria:

* Evidence of a personally signed and dated informed consent document indicating that the subject has been informed of all pertinent aspects of the study before any assessment is performed.
* Healthy male participants who, at the time of screening, are between the ages of 21 and 45 years, inclusive.
* Participants who are willing and able to comply with scheduled visits, treatment plan, bio-imaging procedure, laboratory tests and other study procedures.
* Healthy participant which is defined as in general good physical health, as judged by the investigator and no clinically relevant abnormalities identified by a detailed medical history, full physical examination, including blood pressure and pulse rate measurement, 12-lead Electrocardiogram (ECG) or clinical laboratory tests.
* Body Mass Index (BMI) of 17.5 to 30.5 kilogram per meter square (kg/m2); and a total body weight >50 kg (110 lbs)

Exclusion Criteria:

* Participants who are investigational site staff members directly involved in the conduct of the study and their family members, site staff members otherwise supervised by the investigator, or participants who are GSK employees directly involved in the conduct of the study.
* Participation in other studies involving investigational drug(s) within 30 days prior to study entry and/or during study participation.
* Acute or chronic medical or psychiatric condition or laboratory abnormality that may increase the risk associated with study participation or investigational product administration or may interfere with the interpretation of study results and, in the judgment of the investigator, would make the participant inappropriate for entry into this study.
* Known or suspected intolerance or hypersensitivity or contraindication to the study materials (or closely related compounds) or any of their stated ingredients.
* Participant with known allergy or intolerance to any of the contents of the standard meals.
* Participant is vegetarian.
* Unwilling or unable to comply with the Lifestyle guidelines described in this protocol.
* Use of prescription or non-prescription drugs and dietary supplements within 14 days or 5 half-lives, whichever is longer, prior to the first dose of investigational product that are deemed by the investigator to have a potential impact on the study objectives results.
* Evidence or history of clinically significant laboratory abnormality, hematological, renal, endocrine, pulmonary, cardiovascular, hepatic, psychiatric, neurologic, or allergic disease within the last 5 years that may increase the risk associated with study participation.
* A positive urine drug screen, breath alcohol test or urine cotinine test during Screening or on Day -1 of the study.
* Any condition possibly affecting drug absorption (e.g., gastrectomy)
* A history of current or relevant previous non-self-limiting gastrointestinal disorders peptic ulcer disease and/or gastrointestinal bleeding.
* Currently suffering from disease known to impact gastric emptying, e.g. migraine, insulin-dependent diabetes mellitus.
* The participant has had radiation exposure from clinical trials, including from the present study, and from therapeutic or diagnostic exposure, but excluding background radiation, exceeding a target organ (colon) dose of 50 mSv (5 rems) from a single dose within the last 30 days or a cumulative dose of 150 mSv (15 rems) in the last 12 months. No participant whose occupation requires monitoring for radiation exposure will be enrolled in the study.
* Participants who have been exposed to ionising radiation in excess of 10 mSv (whole body effective dose) above background over the previous 3 years period as a result of occupational exposure or previous participation in research studies. Clinically justified (therapeutic or diagnostic) exposures are not included in this calculation.
* Renal disease or impaired renal function at screening as indicated by abnormal levels of serum creatinine or urea or the presence of clinically significant abnormal urinary constituents (e.g. albuminuria). Minor deviations of laboratory values from the normal range are permitted, if judged by the investigator to have no clinical relevance.
* History or current evidence of ongoing hepatic disease or impaired hepatic function at screening. A candidate will be excluded if more than one of the following lab value deviations are found: 1) AST/SGOT (≥ 1.2 ULN), ALT/SGPT (≥ 1.2 ULN), 2) GGT (≥ 1.2 ULN), ALP (≥ 1.2 ULN), 3) total bilirubin (≥ 1.2 mg/dL) Minor deviations of laboratory values from the normal range are permitted, if judged by the investigator to have no clinical relevance. Positive results in any of the virology tests for HIV-Ab, HCV-Ab, HBsAg and HBc-Ab (Total).
* Diagnosis of long QT syndrome or QTc > 450 msec for males at screening.
* Participants who were intending to father a child in the 3 months following the study.
* Participants who were unwilling to follow contraception requirements
* Participant had any non-removable metal objects such as metal plates, screws etc. in their chest or abdominal area.
* History of regular alcohol consumption exceeding 14 drinks/week (1 drink = 5 ounces (150 mL) of wine or 12 ounces (360 mL) of beer or 1.5 ounces (45 mL) of hard liquor) within 6 months of Screening.
* Smokers defined as the use of tobacco products (including but not limited to: electronic-cigarettes, nicotine gums, nicotine lozenges, etc) during the 6 months prior to screening or a positive urine cotinine test at screening.
* Participant has consumed (eat or drink) grapefruit or grapefruit-related citrus fruits (e.g., Seville oranges, pomelos, pawpaw, dragon fruit, kiwi fruit, mango, passion fruit, pomegranate, rambutan, star fruit or products that contain these fruits) 14 days prior to the first dose of investigational product.
* Participants who have previously been enrolled in this study.

Ages: 21 Years to 45 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 28 (Actual)
Dates: Start 2018-03-01 (Actual); Primary Completion 2018-03-29 (Actual); Study Completion 2018-03-29 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline; GSK Clinical Trials, Study Director — GlaxoSmithKline (for GlaxoSmithKline; Human Genome Sciences Inc., a GSK Company; Sirtris, a GSK Company; Stiefel, a GSK Company; ViiV Healthcare)
Locations (1):
- GSK Investigational Site, Lexington, Kentucky, United States

REFERENCES:
- [Derived] Mallefet P, Armogida M, Doll WJ, Page RC, Sandefer EP. A single-dose, open-label, randomized, scintigraphic study to investigate the gastrointestinal behavior of 2 triple-combination cold products (acetaminophen, phenylephrine, and dextromethorphan) in healthy male volunteers. Trials. 2022 Feb 8;23(1):128. doi: 10.1186/s13063-022-06037-x. PMID 35135601

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were recruited from one center in USA.
Pre-assignment Details: A total of 32 participants were screened, of whom 28 were randomized for treatment and 4 were screen failures.
Groups:
- Treatment Group A: Participants received single oral dose; 1 sachet of Theraflu Daytime Severe Cold and Cough radiolabeled powder (that contained Acetaminophen 650 milligrams [mg] + Phenylephrine 10 mg + Dextromethorphan 20 mg) for oral solution reconstituted with 225 milliliters (mL) of hot water. Participants were instructed to consume the hot drink entirely within 30 seconds on Day 1 morning after an overnight fast and no food or drink was allowed until 4 hours post-dose.
- Treatment Group B: Participants received single oral dose; 2 radiolabeled caplets of Theraflu ExpressMax Daytime Severe Cold and Cough (each caplet contained Acetaminophen 325 mg + Phenylephrine 5 mg + Dextromethorphan 10 mg) with 225 mL of room temperature non-carbonated water. Participants were instructed to consume all the water (225 mL) within 30 seconds on Day 1 morning after an overnight fast and no food or drink was allowed until 4 hours post-dose.
Period: Overall Study
Arm/Group | Treatment Group A | Treatment Group B
Started | 14 | 14
Completed | 14 | 14
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Population: Safety population was defined as all participants who received a radiolabeled treatment A or B irrespective of whether the participant was included in the scintigraphy analysis.
Groups:
- Treatment Group A: Participants received single oral dose; 1 sachet of Theraflu Daytime Severe Cold and Cough radiolabeled powder (that contained Acetaminophen 650 mg + Phenylephrine 10 mg + Dextromethorphan 20 mg) for oral solution reconstituted with 225 mL of hot water. Participants were instructed to consume the hot drink entirely within 30 seconds on Day 1 morning after an overnight fast and no food or drink was allowed until 4 hours post-dose.
- Total: Total of all reporting groups
Arm/Group | Treatment Group A | Treatment Group B | Total
Number analyzed (Participants) | 14 | 14 | 28
Age, Continuous [Mean (Standard Deviation); unit: Years] | 28.0 (8.74) | 28.8 (5.19) | 28.4 (7.06)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 0 | 0
  Male | 14 | 14 | 28
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Height [Mean (Standard Deviation); unit: Centimeters] | 183.1 (6.53) | 180.6 (7.00) | 181.9 (6.76)

OUTCOME MEASURES:

1. Primary Outcome: Mean Time to Onset of Gastric Emptying
Description: Mean time to onset of gastric emptying in participants who did not vomit shortly (within 60 minutes) after study drug administration was evaluated by scintigraphic imaging, performed immediately after ingestion of the investigational drug formulation (radiolabeled with not more than 108 microcurie [mcCi] isotope-technetium-99m-diethylene-triamine-pentaacetate [DTPA]). Data images were analyzed in a time-lapse format and corrected for radioactive decay and background radiation. Regions of interest (ROI) included the stomach, proximal small intestine, distal small intestine and colon.
Time Frame: Predose until 10 hours post dose on Day 1
Population: Scintigraphy analysis population included all participants who received the radiolabeled treatments A or B and who did not vomit shortly (within 60 minutes) after study drug administration, who had sufficient data to determine time to onset and completion of gastric emptying and who had no major protocol deviations.
Measure: Mean (Standard Deviation); unit: minutes
Arm/Group | Treatment Group A | Treatment Group B
Number analyzed (Participants) | 14 | 14
minutes | 1.107 (1.2130) | 8.534 (6.6062)

2. Primary Outcome: Mean Time to Complete Gastric Emptying
Description: Mean time to complete gastric emptying in participants who did not vomit shortly (within 60 minutes) after study drug administration was evaluated by scintigraphic imaging, performed immediately after ingestion of the investigational drug formulation (radiolabeled with not more than 108 mcCi isotope-technetium-99m-DTPA). Data images were analyzed in a time-lapse format and corrected for radioactive decay and background radiation. ROI included the stomach, proximal small intestine, distal small intestine and colon.
Time Frame: Predose until 10 hours post dose on Day 1
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: minutes
Arm/Group | Treatment Group A | Treatment Group B
Number analyzed (Participants) | 14 | 14
minutes | 121.2 (47.76) | 65.3 (47.40)

3. Primary Outcome: Mean Time for Gastric Emptying by Measuring 25 Percent Values
Description: Mean time to gastric emptying by 25 percent (GE25%) was evaluated by scintigraphic imaging, performed immediately after ingestion of the investigational drug formulation (radiolabeled with not more than 108 mcCi isotope-technetium-99m DTPA). Data images were analyzed in a time-lapse format and corrected for radioactive decay and background radiation. ROI included the stomach, proximal small intestine, distal small intestine and colon.
Time Frame: Predose until 10 hours post dose on Day 1
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: minutes
Arm/Group | Treatment Group A | Treatment Group B
Number analyzed (Participants) | 14 | 14
minutes | 12.614 (6.8249) | 12.171 (9.1819)

4. Primary Outcome: Mean Time for Gastric Emptying by Measuring 50 Percent Values
Description: Mean time to gastric emptying by 50 percent (GE50%) was evaluated by scintigraphic imaging, performed immediately after ingestion of the investigational drug formulation (radiolabeled with not more than 108 mcCi isotope-technetium-99m DTPA). Data images were analyzed in a time-lapse format and corrected for radioactive decay and background radiation. ROI included the stomach, proximal small intestine, distal small intestine and colon.
Time Frame: Predose until 10 hours post dose on Day 1
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: minutes
Arm/Group | Treatment Group A | Treatment Group B
Number analyzed (Participants) | 14 | 14
minutes | 22.643 (11.4058) | 16.134 (11.8721)

5. Primary Outcome: Mean Time for Gastric Emptying by Measuring 90 Percent Values
Description: Mean time to gastric emptying by 90 percent (GE90%) was evaluated by scintigraphic imaging, performed immediately after ingestion of the investigational drug formulation (radiolabeled with not more than 108 mcCi isotope-technetium-99m DTPA). Data images were analyzed in a time-lapse format and corrected for radioactive decay and background radiation. ROI included the stomach, proximal small intestine, distal small intestine and colon.
Time Frame: Predose until 10 hours post dose on Day 1
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: minutes
Arm/Group | Treatment Group A | Treatment Group B
Number analyzed (Participants) | 14 | 14
minutes | 84.929 (43.1606) | 36.214 (33.7711)

6. Primary Outcome: Percentage of Radiolabeled Drug Remaining in the Stomach After 15 Minutes of Administration
Description: Percentage of radiolabeled drug remaining in the stomach was evaluated by scintigraphic imaging, performed immediately after ingestion of the investigational drug formulation (radiolabeled with not more than 108 mcCi isotope-technetium-99m DTPA) and after 15 minutes of drug ingestion. Data images were analyzed and corrected for radioactive decay and background radiation.
Time Frame: 15 minutes post dose on Day 1
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: percentage of radiolabeled drug
Arm/Group | Treatment Group A | Treatment Group B
Number analyzed (Participants) | 14 | 14
percentage of radiolabeled drug | 67.00 (13.260) | 49.77 (42.193)

7. Primary Outcome: Percentage of Radiolabeled Drug Remaining in the Stomach After 30 Minutes of Administration
Description: Percentage of radiolabeled drug remaining in the stomach was evaluated by scintigraphic imaging, performed immediately after ingestion of the investigational drug formulation (radiolabeled with not more than 108 mcCi isotope-technetium-99m DTPA) and after 30 minutes of drug ingestion. Data images were analyzed and corrected for radioactive decay and background radiation.
Time Frame: 30 minutes post dose on Day 1
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: percentage of radiolabeled drug
Arm/Group | Treatment Group A | Treatment Group B
Number analyzed (Participants) | 14 | 14
percentage of radiolabeled drug | 33.24 (19.321) | 20.87 (26.697)

8. Primary Outcome: Percentage of Radiolabeled Drug Remaining in the Stomach After 45 Minutes of Administration
Description: Percentage of radiolabeled drug remaining in the stomach was evaluated by scintigraphic imaging, performed immediately after ingestion of the investigational drug formulation (radiolabeled with not more than 108 mcCi isotope-technetium-99m DTPA) and after 45 minutes of drug ingestion. Data images were analyzed and corrected for radioactive decay and background radiation.
Time Frame: 45 minutes post dose on Day 1
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: percentage of radiolabeled drug
Arm/Group | Treatment Group A | Treatment Group B
Number analyzed (Participants) | 14 | 14
percentage of radiolabeled drug | 24.79 (16.334) | 7.21 (11.387)

9. Primary Outcome: Percentage of Radiolabeled Drug Remaining in the Stomach After 60 Minutes of Administration
Description: Percentage of radiolabeled drug remaining in the stomach was evaluated by scintigraphic imaging, performed immediately after ingestion of the investigational drug formulation (radiolabeled with not more than 108 mcCi isotope-technetium-99m DTPA) and after 60 minutes of drug ingestion. Data images were analyzed and corrected for radioactive decay and background radiation.
Time Frame: 60 minutes post dose on Day 1
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: percentage of radiolabeled drug
Arm/Group | Treatment Group A | Treatment Group B
Number analyzed (Participants) | 14 | 14
percentage of radiolabeled drug | 20.07 (13.885) | 4.26 (10.378)

10. Primary Outcome: Percentage of Radiolabeled Drug Remaining in the Stomach After 75 Minutes of Administration
Description: Percentage of radiolabeled drug remaining in the stomach was evaluated by scintigraphic imaging, performed immediately after ingestion of the investigational drug formulation (radiolabeled with not more than 108 mcCi isotope-technetium-99m DTPA) and after 75 minutes of drug ingestion. Data images were analyzed and corrected for radioactive decay and background radiation.
Time Frame: 75 minutes post dose on Day 1
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: percentage of radiolabeled drug
Arm/Group | Treatment Group A | Treatment Group B
Number analyzed (Participants) | 14 | 14
percentage of radiolabeled drug | 14.73 (13.350) | 3.28 (8.123)

11. Primary Outcome: Percentage of Radiolabeled Drug Remaining in the Stomach After 90 Minutes of Administration
Description: Percentage of radiolabeled drug remaining in the stomach was evaluated by scintigraphic imaging, performed immediately after ingestion of the investigational drug formulation (radiolabeled with not more than 108 mcCi isotope-technetium-99m DTPA) and after 90 minutes of drug ingestion. Data images were analyzed and corrected for radioactive decay and background radiation.
Time Frame: 90 minutes post dose on Day 1
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: percentage of radiolabeled drug
Arm/Group | Treatment Group A | Treatment Group B
Number analyzed (Participants) | 14 | 14
percentage of radiolabeled drug | 8.84 (9.867) | 2.45 (6.164)

12. Primary Outcome: Percentage of Radiolabeled Drug Remaining in the Stomach After 105 Minutes of Administration
Description: Percentage of radiolabeled drug remaining in the stomach was evaluated by scintigraphic imaging, performed immediately after ingestion of the investigational drug formulation (radiolabeled with not more than 108 mcCi isotope-technetium-99m DTPA) and after 105 minutes of drug ingestion. Data images were analyzed and corrected for radioactive decay and background radiation.
Time Frame: 105 minutes post dose on Day 1
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: percentage of radiolabeled drug
Arm/Group | Treatment Group A | Treatment Group B
Number analyzed (Participants) | 14 | 14
percentage of radiolabeled drug | 6.06 (8.145) | 1.72 (5.279)

13. Primary Outcome: Percentage of Radiolabeled Drug Remaining in the Stomach After 120 Minutes of Administration
Description: Percentage of radiolabeled drug remaining in the stomach was evaluated by scintigraphic imaging, performed immediately after ingestion of the investigational drug formulation (radiolabeled with not more than 108 mcCi isotope-technetium-99m DTPA) and after 120 minutes of drug ingestion. Data images were analyzed and corrected for radioactive decay and background radiation.
Time Frame: 120 minutes post dose on Day 1
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: percentage of radiolabeled drug
Arm/Group | Treatment Group A | Treatment Group B
Number analyzed (Participants) | 14 | 14
percentage of radiolabeled drug | 4.34 (6.177) | 0.99 (3.546)

14. Primary Outcome: Percentage of Radiolabeled Drug Remaining in the Stomach After 180 Minutes of Administration
Description: Percentage of radiolabeled drug remaining in the stomach was evaluated by scintigraphic imaging, performed immediately after ingestion of the investigational drug formulation (radiolabeled with not more than 108 mcCi isotope-technetium-99m DTPA) and after 180 minutes of drug ingestion. Data images were analyzed and corrected for radioactive decay and background radiation.
Time Frame: 180 minutes post dose on Day 1
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: percentage of radiolabeled drug
Arm/Group | Treatment Group A | Treatment Group B
Number analyzed (Participants) | 14 | 14
percentage of radiolabeled drug | 0.64 (2.108) | 0.00 (0.000)

15. Primary Outcome: Percentage of Radiolabeled Drug Remaining in the Stomach After 240 Minutes of Administration
Description: Percentage of radiolabeled drug remaining in the stomach was evaluated by scintigraphic imaging, performed immediately after ingestion of the investigational drug formulation (radiolabeled with not more than 108 mcCi isotope-technetium-99m DTPA) and after 240 minutes of drug ingestion. Data images were analyzed and corrected for radioactive decay and background radiation.
Time Frame: 240 minutes post dose on Day 1
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: percentage of radiolabeled drug
Arm/Group | Treatment Group A | Treatment Group B
Number analyzed (Participants) | 14 | 14
percentage of radiolabeled drug | 0.00 (0.00) | 0.00 (0.00)

16. Primary Outcome: Area Under the Gastric Emptying Curve From Time 0 to 15 Minutes
Description: Area under the gastric emptying curve from time 0 to 15 was evaluated by scintigraphic imaging, performed immediately after ingestion of the investigational drug formulation (radiolabeled with not more than 108 mcCi isotope-technetium-99m DTPA) and after 15 minutes of drug ingestion. Data images were analyzed and corrected for radioactive decay and background radiation.
Time Frame: 15 minutes post dose on Day 1
Population: as for outcome 1
Measure: Mean (Standard Error); unit: percentage dose*hour
Arm/Group | Treatment Group A | Treatment Group B
Number analyzed (Participants) | 14 | 14
percentage dose*hour | 19.38 (0.511) | 16.96 (1.769)

17. Primary Outcome: Area Under the Gastric Emptying Curve From Time 0 to 30 Minutes
Description: Area under the gastric emptying curve from time 0 to 30 was evaluated by scintigraphic imaging, performed immediately after ingestion of the investigational drug formulation (radiolabeled with not more than 108 mcCi isotope-technetium-99m DTPA) and after 30 minutes of drug ingestion. Data images were analyzed and corrected for radioactive decay and background radiation.
Time Frame: 30 minutes post dose on Day 1
Population: as for outcome 1
Measure: Mean (Standard Error); unit: percentage dose*hour
Arm/Group | Treatment Group A | Treatment Group B
Number analyzed (Participants) | 14 | 14
percentage dose*hour | 31.16 (1.598) | 25.11 (3.873)

18. Primary Outcome: Area Under the Gastric Emptying Curve From Time 0 to 45 Minutes
Description: Area under the gastric emptying curve from time 0 to 45 was evaluated by scintigraphic imaging, performed immediately after ingestion of the investigational drug formulation (radiolabeled with not more than 108 mcCi isotope-technetium-99m DTPA) and after 45 minutes of drug ingestion. Data images were analyzed and corrected for radioactive decay and background radiation.
Time Frame: 45 minutes post dose on Day 1
Population: as for outcome 1
Measure: Mean (Standard Error); unit: percentage dose*hour
Arm/Group | Treatment Group A | Treatment Group B
Number analyzed (Participants) | 14 | 14
percentage dose*hour | 38.36 (2.727) | 28.19 (4.864)

19. Primary Outcome: Area Under the Gastric Emptying Curve From Time 0 to 60 Minutes
Description: Area under the gastric emptying curve from time 0 to 60 was evaluated by scintigraphic imaging, performed immediately after ingestion of the investigational drug formulation (radiolabeled with not more than 108 mcCi isotope-technetium-99m DTPA) and after 60 minutes of drug ingestion. Data images were analyzed and corrected for radioactive decay and background radiation.
Time Frame: 60 minutes post dose on Day 1
Population: as for outcome 1
Measure: Mean (Standard Error); unit: percentage dose*hour
Arm/Group | Treatment Group A | Treatment Group B
Number analyzed (Participants) | 14 | 14
percentage dose*hour | 43.69 (3.620) | 29.60 (5.402)

20. Primary Outcome: Area Under the Gastric Emptying Curve From Time 0 to 75 Minutes
Description: Area under the gastric emptying curve from time 0 to 75 was evaluated by scintigraphic imaging, performed immediately after ingestion of the investigational drug formulation (radiolabeled with not more than 108 mcCi isotope-technetium-99m DTPA) and after 75 minutes of drug ingestion. Data images were analyzed and corrected for radioactive decay and background radiation.
Time Frame: 75 minutes post dose on Day 1
Population: as for outcome 1
Measure: Mean (Standard Error); unit: percentage dose*hour
Arm/Group | Treatment Group A | Treatment Group B
Number analyzed (Participants) | 14 | 14
percentage dose*hour | 48.71 (4.659) | 30.61 (5.888)

21. Primary Outcome: Area Under the Gastric Emptying Curve From Time 0 to 90 Minutes
Description: Area under the gastric emptying curve from time 0 to 90 was evaluated by scintigraphic imaging, performed immediately after ingestion of the investigational drug formulation (radiolabeled with not more than 108 mcCi isotope-technetium-99m DTPA) and after 90 minutes of drug ingestion. Data images were analyzed and corrected for radioactive decay and background radiation.
Time Frame: 90 minutes post dose on Day 1
Population: as for outcome 1
Measure: Mean (Standard Error); unit: percentage dose*hour
Arm/Group | Treatment Group A | Treatment Group B
Number analyzed (Participants) | 14 | 14
percentage dose*hour | 51.32 (5.242) | 31.29 (6.236)

22. Primary Outcome: Area Under the Gastric Emptying Curve From Time 0 to 105 Minutes
Description: Area under the gastric emptying curve from time 0 to 105 was evaluated by scintigraphic imaging, performed immediately after ingestion of the investigational drug formulation (radiolabeled with not more than 108 mcCi isotope-technetium-99m DTPA) and after 105 minutes of drug ingestion. Data images were analyzed and corrected for radioactive decay and background radiation.
Time Frame: 105 minutes post dose on Day 1
Population: as for outcome 1
Measure: Mean (Standard Error); unit: percentage dose*hour
Arm/Group | Treatment Group A | Treatment Group B
Number analyzed (Participants) | 14 | 14
percentage dose*hour | 53.16 (5.745) | 31.81 (6.529)

23. Primary Outcome: Area Under the Gastric Emptying Curve From Time 0 to 120 Minutes
Description: Area under the gastric emptying curve from time 0 to 120 was evaluated by scintigraphic imaging, performed immediately after ingestion of the investigational drug formulation (radiolabeled with not more than 108 mcCi isotope-technetium-99m DTPA) and after 120 minutes of drug ingestion. Data images were analyzed and corrected for radioactive decay and background radiation.
Time Frame: 120 minutes post dose on Day 1
Population: as for outcome 1
Measure: Mean (Standard Error); unit: percentage dose*hour
Arm/Group | Treatment Group A | Treatment Group B
Number analyzed (Participants) | 14 | 14
percentage dose*hour | 54.49 (6.138) | 32.15 (6.743)

24. Primary Outcome: Area Under the Gastric Emptying Curve From Time 0 to 180 Minutes
Description: Area under the gastric emptying curve from time 0 to 180 was evaluated by scintigraphic imaging, performed immediately after ingestion of the investigational drug formulation (radiolabeled with not more than 108 mcCi isotope-technetium-99m DTPA) and after 180 minutes of drug ingestion. Data images were analyzed and corrected for radioactive decay and background radiation.
Time Frame: 180 minutes post dose on Day 1
Population: as for outcome 1
Measure: Mean (Standard Error); unit: percentage dose*hour
Arm/Group | Treatment Group A | Treatment Group B
Number analyzed (Participants) | 14 | 14
percentage dose*hour | 56.69 (6.992) | 32.61 (7.069)

25. Primary Outcome: Area Under the Gastric Emptying Curve From Time 0 to 240 Minutes
Description: Area under the gastric emptying curve from time 0 to 240 was evaluated by scintigraphic imaging, performed immediately after ingestion of the investigational drug formulation (radiolabeled with not more than 108 mcCi isotope-technetium-99m DTPA) and after 240 minutes of drug ingestion. Data images were analyzed and corrected for radioactive decay and background radiation.
Time Frame: 240 minutes post dose on Day 1
Population: as for outcome 1
Measure: Mean (Standard Error); unit: percentage dose*hour
Arm/Group | Treatment Group A | Treatment Group B
Number analyzed (Participants) | 14 | 14
percentage dose*hour | 56.80 (7.071) | 32.61 (7.069)

26. Primary Outcome: Total Area Under the Gastric Emptying Curve
Description: Total area under the gastric emptying curve was evaluated by scintigraphic imaging, performed after ingestion of the investigational drug formulation (radiolabeled with not more than 108 mcCi isotope-technetium-99m DTPA). Data images were analyzed in a time-lapse format and corrected for radioactive decay and background radiation.
Time Frame: Predose until 10 hours post dose on Day 1
Population: as for outcome 1
Measure: Mean (Standard Error); unit: percentage dose*hour
Arm/Group | Treatment Group A | Treatment Group B
Number analyzed (Participants) | 14 | 14
percentage dose*hour | 56.80 (7.071) | 32.61 (7.069)

27. Primary Outcome: Gastric Emptying Half-Life
Description: Gastric emptying half-life was defined as the time required by the stomach to empty 50% of the ingested meal and was evaluated by scintigraphic imaging, performed immediately after ingestion of the investigational drug formulation (radiolabeled with not more than 108 mcCi isotope-technetium-99m DTPA). Data images were analyzed in a time-lapse format and corrected for radioactive decay and background radiation.
Time Frame: Predose until 10 hours post dose on Day 1
Population: as for outcome 1
Measure: Median (Full Range); unit: minutes
Arm/Group | Treatment Group A | Treatment Group B
Number analyzed (Participants) | 14 | 14
minutes | 25.00 [6.8 to 52.0] | 5.00 [1.0 to 35.0]

28. Primary Outcome: Small Intestine Transit Time
Description: Small intestinal transit time was calculated by determining the arrival time of the radiolabeled investigational drug formulation at the cecum or colon region from scintigraphic imaging and subtracting the gastric emptying value.
Time Frame: Predose until 10 hours post dose on Day 1
Population: as for outcome 1
Measure: Median (Full Range); unit: minutes
Arm/Group | Treatment Group A | Treatment Group B
Number analyzed (Participants) | 14 | 14
minutes | 184.0 [106 to 265] | 139.5 [61 to 243]

29. Secondary Outcome: Number of Participants With Clinically Significant Change in Laboratory Test Values
Description: Haematological, biochemistry, urinalysis and virological parameters were analyzed. Clinical significance was judged by the investigator based upon the out of range values of standard range set for each parameter.
Time Frame: From baseline up to Day 1
Population: as for baseline characteristics
Measure: Count of Participants; unit: Participants
Arm/Group | Treatment Group A | Treatment Group B
Number analyzed (Participants) | 14 | 14
Participants | 0 | 0

ADVERSE EVENTS:
Time Frame: From signature of informed consent form up to 5 days after last administration of the investigational product (up to Day 6)
Description: Safety population was defined as all participants who received a radiolabeled treatment A or B irrespective of whether the participant was included in the scintigraphy analysis. All AEs were summarized by system organ class and preferred term. All treatment emergent AEs and SAEs were collected and reported.
Arm/Group | Treatment Group A | Treatment Group B
All-Cause Mortality (participants affected / at risk) | 0/14 | 0/14
Serious Adverse Events (participants affected / at risk) | 0/14 | 0/14
Other Adverse Events (participants affected / at risk) | 1/14 | 2/14
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Treatment Group A (N=14) | Treatment Group B (N=14)
Diarrhoea (Gastrointestinal disorders) | 0 (0) | 1 (1)
Nausea (Gastrointestinal disorders) | 0 (0) | 1 (1)
Fatigue (General disorders) | 1 (1) | 0 (0)
Alanine aminotransferase increased (Investigations) | 0 (0) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
GSK agreements may vary with individual investigators but will not prohibit any investigator from publishing. GSK supports the publication of results from all centers of a multi-center trial but requests that reports based on single-site data not precede the primary publication of the entire clinical trial.

DOCUMENTS (2):
  • Study Protocol (2018-01-25): https://cdn.clinicaltrials.gov/large-docs/43/NCT03415243/Prot_000.pdf
  • Statistical Analysis Plan (2018-02-27): https://cdn.clinicaltrials.gov/large-docs/43/NCT03415243/SAP_001.pdf